CLINICAL TRIAL: NCT06136637
Title: Evaluation de l'utilité du Monitorage du Glycacalyx Pour prédire Les Complications du Patient de Chirurgie Cardiaque
Brief Title: Monitoring of Glycocalyx for Prediction of Complications After Cardiac Surgery
Acronym: MOGLYCC
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Collaborators: University of Rouen Normandie (Other)
Responsible Party: Principal Investigator, DEMAILLY Zoe, Principal Investigator, University Hospital, Rouen
Other Study IDs: 2021-A02377-34; 2020/416/OB (Other: DRCI CHU Rouen)
Record Dates: First submitted 2023-03-29; First posted 2023-11-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Cardiac Surgery
Keywords: Glycocalyx; Microcirculation; Cardiopulmonary bypass; Organ failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective observational study of the evolution of the microcirculation and the sublingual glycocalyx in perioperative cardiac surgery under cardiopulmonary bypass. Our main objective is to evaluate the prognostic value of the variation of the thickness of the perioperative glycocalyx for the occurrence of a major complication in the first 24 hours after surgery.

ELIGIBILITY:
* Patient of legal age (age ≥ 18 years)
* Patient undergoing scheduled cardiac surgery with cardiopulmoary bypass (CPB) (expected duration of CPB > 60 min)
* Person informed with collection of non-opposition at the latest, the day before the operation - Person affiliated to a social security system

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient undergoing cardiac surgery with cardiopulmonary bypass
Sampling Method: Non-Probability Sample
Enrollment: 77 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Glycocalyx thickness variation | Two hours after the end of cardiopulmonarybypass
  Change in glycocalyx thickness between the preoperative period and the postoperative period (2 hours after the end of cardiopulmonary bypass).

CONTACTS AND LOCATIONS:
Locations (1):
- Rouen University Hospital, Rouen, France